CLINICAL TRIAL: NCT01120652
Title: Reducing Depressive Symptoms in Systemic Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Carol Greco, Assistant Professor of Psychiatry, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR057338
Record Dates: First submitted 2010-04-08; First posted 2010-05-11 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Skills Training (Experimental): This is a behavioral intervention that blends cognitive-behavioral therapy methods, mind-body relaxation training, and mindfulness practices.
  Interventions: Behavioral: Mind-Body Skills Training (MBST)
- Supportive Counseling (Active Comparator): This is a behavioral intervention consisting of support and symptom monitoring but without specific skills training or provision of advice.
  Interventions: Behavioral: Supportive Counseling (SC)

INTERVENTIONS:
Behavioral: Mind-Body Skills Training (MBST) — This is a behavioral intervention that blends cognitive-behavioral therapy methods, mind-body relaxation training, and mindfulness practices. MBST is provided in 8 individual sessions, each lasting approximately one hour. Ideally, sessions take place on a weekly basis, so that the intervention phase of the study lasts for approximately two months.
  Arms: Mind-Body Skills Training
Behavioral: Supportive Counseling (SC) — This is a behavioral intervention consisting of support and symptom monitoring but without specific skills training or provision of advice. SC is provided in 8 individual sessions, each lasting approximately one hour. Ideally, sessions take place on a weekly basis, so that the intervention phase of the study lasts for approximately two months.
  Arms: Supportive Counseling

SUMMARY:
The purpose of this randomized controlled trial is to evaluate the efficacy of a Mind-Body Skills Training intervention for improving mental and physical health in patients with Systemic Lupus Erythematosus (SLE) who have comorbid depressive symptoms.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic, multisystemic inflammatory disease that is frequently associated with significant psychological suffering. Building upon our team's strengths in lupus biomedical research and behavioral interventions, we propose to study a non-pharmacologic intervention to improve mental and physical health of patients with SLE and co-morbid depression.

In this project, entitled, Reducing Depressive Symptoms in SLE, we will investigate the efficacy of an innovative non-pharmacologic intervention, Mind-Body Skills Training (MBST) for improving mental and physical health outcomes in SLE in a randomized controlled trial (RCT). MBST is a novel approach that combines cognitive-behavioral therapy methods, mind-body relaxation skills, and mindfulness components, each of which is beneficial for reducing pain and/or distress in other inflammatory conditions. We will assign 150 SLE patients with depressive disorder or subsyndromal depression to MBST or to a supportive counseling control condition. The primary specific aims of the project are to evaluate the effects of the 8-session MBST program on 1) mental health (depression) and 2) physical health (pain, fatigue, and health-related quality of life). Additionally we will explore the effects of the MBST intervention on 1) novel SLE biomarkers of inflammation and immune function: cell-bound complement activation products, developed at our site, 2) measures of SLE disease activity, and we will explore 3) potential treatment modifiers and mediators: baseline pain and socioeconomic status, and self-efficacy and perceived stress. We will evaluate health outcomes after the interventions and at 6- and 12-months follow-up.

SLE is one of the most complex autoimmune diseases, with one of the highest rates of depression. The MBST intervention has strong potential for addressing the unique physical manifestations and mental suffering in this patient group, and may have broad impact on distressed patients with other debilitating chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE according to 1997 updated SLE criteria (Hochberg 1997)
* Women and men of all races/ethnic groups age 18 and over
* Able to speak and read English
* Willing to be randomized to either MBST or SC and attend sessions
* Medications stable for at least one month
* Dose of prednisone or equivalent < 15 mg per day
* PHQ-9 score > or = 9
* BILAG classification B, C, D, or E: indicating a level of SLE activity not requiring new or increased medication
* CES-D score > or = 16
* QIDS-C endorsement of subsyndromal or greater depression symptoms
* Not currently seeking psychiatric disability benefits

Exclusion Criteria:

* BILAG A, indicating new SLE flare requiring an immediate dose adjustment or addition of corticosteroid or immunosuppressant treatment.
* Uncontrolled medical condition (e.g., severe infection) that is determined by the research physicians to put the participant at undue risk or to interfere with ability to participate in the study.
* Psychosis, bipolar disorder, actively suicidal or otherwise requiring immediate psychiatric treatment, as determined by diagnostic interview (SCID).
* Current skills-based psychotherapy. However, if patients are currently receiving supportive psychotherapy and are willing to suspend this for the duration of the intervention period, they may enroll in the study.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression scale (CESD) | approximately 1 year following the 8 session intervention
  The CESD is a self report questionnaire designed to assess depressive symptoms.

SECONDARY OUTCOMES:
Pain (Multidimensional Pain Inventory - Pain Severity scale) | approximately 1 year following the 8 session intervention
  The MPI Pain Severity scale is a 3 item self report instrument to assess current and past week pain severity
Fatigue (PROMIS - fatigue scale - short form) | approximately 1 year following the 8 session intervention
  The Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue short form scale assesses past week fatigue.
Health-related quality of life (SF-12 health survey) | approximately 1 year following the 8 session intervention

CONTACTS AND LOCATIONS:
Overall Officials: Carol M. Greco, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States